CLINICAL TRIAL: NCT00425308
Title: A Prospective Multicenter Open-label Randomized Study to Assess Efficacy and Safety of Everolimus in Combination With Cyclosporine Microemulsion Versus Everolimus Without Calcineurine Inhibitor in Combination With Enteric-coated Mycophenolate Sodium (EC-MPS), in Adult Renal Transplant Patients in Maintenance.
Brief Title: Efficacy and Safety of Everolimus in Combination With Cyclosporine Microemulsion Versus Everolimus in Combination With Enteric-coated Mycophenolate Sodium (EC-MPS), in Adult Renal Transplant Patients in Maintenance.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AFR06
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
Keywords: Everolimus, calcineurine inhibitor, renal transplantation in maintenance, chronic allograft nephropathy
MeSH Terms: interventions — Everolimus; Cyclosporine; Mycophenolic Acid; Steroids

ARMS (2):
- Everolimus + Enteric-coated Mycophenolate Sodium (EC-MPS) (Active Comparator): Everolimus dose has been adjusted to reach in Group 2, assessment of everolimus dose/trough level (C0), between 6 and 10 ng/ml plus Enteric-coated Mycophenolate Sodium (EC-MPS) 720 mg/d (360mg the morning and 360 mg the evening) plus steroids
  Interventions: Drug: Everolimus + Enteric-coated Mycophenolate Sodium (EC-MPS); Drug: Steroids
- Everolimus + Cyclosporine (Active Comparator): Everolimus dose has been adjusted to reach in Group 1, assessment of everolimus dose/trough level (C0), between 3 and 8 ng/ml plus Cyclosporine in which Group 1 dose adjusted to reach, assessment of Cyclosporine dosage and blood concentration (C2), between 200 and 450 ng/ml plus steroids
  Interventions: Drug: Everolimus + Cyclosporine; Drug: Steroids

INTERVENTIONS:
Drug: Everolimus + Cyclosporine
  Other Names: Cyclosporine Microemulsion; Neoral
  Arms: Everolimus + Cyclosporine
Drug: Everolimus + Enteric-coated Mycophenolate Sodium (EC-MPS)
  Other Names: Myfortic
  Arms: Everolimus + Enteric-coated Mycophenolate Sodium (EC-MPS)
Drug: Steroids

SUMMARY:
Efficacy and safety of 2 groups of treatment: everolimus in association with cyclosporine microemulsion and steroids versus everolimus in association with Enteric-coated Mycophenolate Sodium (EC-MPS) and steroids. The study population consists of patients having taken part in study CRAD001A2420 (NCT00154297) until the end (12 months) and having not prematurely discontinued the immunosuppressive regimen received in this study (everolimus + cyclosporine microemulsion + steroids).

ELIGIBILITY:
Inclusion criteria:

* Patients who participated in and completed study CRAD001A2420

Exclusion criteria:

* Premature study or study treatment discontinuation in CRAD001A2420 study.
* Acute rejection within the 3 months prior to inclusion

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a prospective, national, multicenter, randomized, open label study, 12 months duration. Ten centers have been included with a study start October 2006 and end date May 2009.
Groups:
- Cyclosporine: Control Arm: Everolimus dose has been adjusted to reach in Group 1, assessment of everolimus dose/trough level (C0), between 3 and 8 ng/ml plus Cyclosporine in which Group 1 dose adjusted to reach, assessment of Cyclosporine dosage and blood concentration (C2), between 200 and 450 ng/ml plus steroids
- Enteric-coated Mycophenolate Sodium (EC-MPS): Everolimus dose has been adjusted to reach in Group 2, assessment of everolimus dose/trough level (C0), between 6 and 10 ng/ml plus Enteric-Coated Mycophenolate Sodium (EC-MPS) 720 mg/d (360mg the morning and 360 mg the evening) plus steroids
Period: Overall Study
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Started | 15 | 15
Completed | 11 | 14
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.46) | 58.8 (7.55) | 60.6 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate Estimated by Iohexol Plasma Clearance 12 Months After Randomization Between the 2 Groups of Patients.
Description: Primary efficacy endpoint: between treatment analysis of change in iohexol plasmatic clearance (mL/min) from baseline to Month 12 (M12)
Time Frame: From Baseline to Month 12
Population: Intent to Treat (ITT) Population: all patients with a baseline value
Measure: Least Squares Mean (Standard Error); unit: (mL/min)
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
(mL/min) | -4.07 (5.03) | 10.30 (4.84)

2. Primary Outcome: Change in the Glomerular Filtration Rate Estimated by Iohexol Plasma Clearance 12 Months After Randomization Between the 2 Groups of Patients Who Completed Trial
Description: as for outcome 1
Time Frame: From Baseline to Month 12
Population: Intent to Treat (ITT) Population: completed patients
Measure: Least Squares Mean (Standard Error); unit: (mL/min)
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 8 | 13
(mL/min) | 1.46 (6.60) | 12.00 (5.06)

3. Secondary Outcome: Change in Renal Function Assessed by Serum Creatinine at Month 3, Month 6 and Month 12
Time Frame: From Baseline to Month 3, 6, and 12
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
µmol/L
  Baseline [N = 13; N = 14] | 161.7 (60.78) | 153.2 (47.46)
  Month 3 [N = 12; N = 14] | 156.6 (51.41) | 138.9 (40.85)
  Month 6 [N = 12; N = 13] | 170.8 (59.36) | 139.8 (42.81)
  Month 12 [N = 13; N = 14] | 227.7 (144.0) | 130.4 (40.27)

4. Secondary Outcome: Number of Participants With Biopsy-proven Acute Rejection (BPAR) at Month 6 and Month 12.
Time Frame: Month 6 and 12
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
participants
  Yes: treatment failure Month 6 | 0 | 0
  No: treatment failure Month 6 | 0 | 0
  Yes: treatment failure Month 12 | 1 | 0
  No: treatment failure Month 12 | 12 | 14

5. Secondary Outcome: Number of Participants With Treatment Failures Assessed by Biopsy-proven Acute Rejection (BPAR), Graft Loss/Re-transplantation, Death or Lost to Follow-up at Month 12.
Time Frame: Month 12
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
participants
  BPAR 12 months | 1 | 0
  Graft Loss 12 months | 0 | 0
  Death 12 months | 1 | 0
  Lost to Follow-up 12 months | 0 | 0

6. Secondary Outcome: Change in Renal Function Assessed by Creatinine Clearance at Month 3, Month 6 and Month 12
Description: Change in creatinine clearance, Nankivell formula (mL/min/1.73m²) from baseline to M12
Time Frame: From Baseline to Month 3, 6, and 12
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mL/min/1.73m²
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
mL/min/1.73m²
  Baseline [N = 12; N = 13] | 56.3 (20.07) | 60.3 (18.49)
  Month 3 [N = 10; N = 14] | 57.3 (19.49) | 67.1 (19.24)
  Month 6 [N = 10; N = 12] | 50.3 (15.98) | 68.1 (18.25)
  Month 12 [N = 7; N = 11] | 48.7 (24.70) | 70.1 (18.34)

7. Secondary Outcome: Change in Renal Function Assessed by Proteinuria at Month 3, Month 6 and Month 12
Description: Change in proteinuria (g/24h) from baseline to M12
Time Frame: From Baseline to Month 3, 6, and 12
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: g/24h
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 13 | 14
g/24h
  Baseline [N = 9; N = 10] | 0.44 (0.447) | 0.47 (0.390)
  Month 3 [N = 9; N = 8] | 0.53 (0.248) | 0.24 (0.267)
  Month 6 [N = 6; N = 5] | 0.44 (0.335) | 0.33 (0.262)
  Month 12 [N = 7; N = 10] | 0.48 (0.537) | 0.75 (0.732)

8. Secondary Outcome: Assessing Cardiovascular Risk Factors Based on Fasting Glucose.
Description: Blood chemistry - fasting glycemia (mmol/L)
Time Frame: From Baseline to Month 1, 3, 6, 9, and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 15 | 15
mmol/L
  Baseline [N = 15; N = 15] | 5.5 (0.97) | 5.2 (0.47)
  Month 1 [N = 15; N = 15] | 5.2 (0.90) | 5.3 (0.95)
  Month 3 [N = 14; N = 15] | 5.6 (1.26) | 5.2 (1.26)
  Month 6 [N = 14; N = 14] | 5.5 (1.15) | 5.1 (1.06)
  Month 9 [N = 12; N = 13] | 5.3 (1.04) | 5.6 (1.60)
  Month 12 [N = 14; N = 13] | 4.8 (0.94) | 5.4 (1.21)

9. Secondary Outcome: Assessing Cardiovascular Risk Factors Based on Fasting Total Cholesterol.
Description: Blood chemistry - total cholesterol (mmol/L)
Time Frame: From Baseline to Month 1, 3, 6, 9, and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 15 | 15
mmol/L
  Baseline [N = 13; N = 14] | 5.7 (1.42) | 6.0 (2.26)
  Month 1 [N = 11; N = 14] | 5.0 (1.20) | 5.7 (0.76)
  Month 3 [N = 13; N = 14] | 5.3 (1.77) | 5.6 (1.43)
  Month 6 [N = 12; N = 12] | 5.5 (1.60) | 5.7 (1.78)
  Month 9 [N = 9; N = 12] | 5.4 (1.49) | 5.4 (1.31)
  Month 12 [N = 12; N = 11] | 5.6 (1.61) | 5.8 (0.60)

10. Secondary Outcome: Assessing Cardiovascular Risk Factors Based on Fasting High-density Lipoprotein (HDL) Cholesterol, Low-density Lipoprotein (LDL) Cholesterol.
Time Frame: From Baseline to Month 3, 6, and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 15 | 15
mmol/L
  Baseline LDL [N = 10; N = 14] | 3.4 (0.89) | 3.1 (0.84)
  Baseline HDL [N = 10; N = 14] | 1.5 (0.54) | 1.5 (0.51)
  Month 3 LDL [N = 12; N = 14] | 3.2 (0.89) | 3.4 (0.97)
  Month 3 HDL [N = 12; N = 13] | 1.7 (0.75) | 1.5 (0.37)
  Month 6 LDL [N = 12; N = 12] | 3.2 (1.15) | 3.3 (1.48)
  Month 6 HDL [N = 12; N = 12] | 1.6 (0.47) | 1.4 (0.50)
  Month 12 LDL [N = 10; N = 11] | 3.0 (0.84) | 3.2 (0.65)
  Month 12 HDL [N = 10; N = 11] | 1.7 (0.74) | 1.5 (0.52)

11. Secondary Outcome: Assessing Cardiovascular Risk Factors Based on Fasting Triglycerides.
Time Frame: From Baseline to Month 1, 3, 6, 9, and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 15 | 15
mmol/L
  Baseline [N = 11; N = 14] | 2.4 (1.43) | 1.8 (0.93)
  Month 1 [N = 10; N = 14] | 2.1 (1.16) | 2.0 (0.81)
  Month 3 [N = 13; N = 14] | 2.0 (0.78) | 2.2 (0.78)
  Month 6 [N = 12; N = 12] | 1.9 (0.51) | 2.1 (0.68)
  Month 9 [N = 10; N = 12] | 1.9 (0.77) | 2.2 (0.94)
  Month 12 [N = 12; N = 11] | 2.3 (1.05) | 2.3 (0.95)

12. Secondary Outcome: Assessing Cardiovascular Risk Factors Based on Fasting C-reactive Protein (CRP).
Description: Blood chemistry - C-reactive Protein (CRP) (mg/L)
Time Frame: From Baseline to Month 3, 6, and 12
Population: Safety population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cyclosporine | Enteric-coated Mycophenolate Sodium (EC-MPS)
Number analyzed (Participants) | 15 | 15
mg/L
  Baseline [N = 13; N = 14] | 11.4 (17.83) | 3.0 (2.45)
  Month 3 [N = 11; N = 11] | 6.3 (4.88) | 10.3 (16.27)
  Month 6 [N = 11; N = 9] | 8.0 (8.24) | 5.6 (5.75)
  Month 12 [N = 14; N = 12] | 34.2 (62.92) | 12.6 (27.23)

ADVERSE EVENTS:
Arm/Group | Cyclosporine | Enteric-Coated Mycophenolate Sodium (EC-MPS)
Serious Adverse Events (participants affected / at risk) | 8/15 | 10/15
Other Adverse Events (participants affected / at risk) | 11/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=15) | Enteric-Coated Mycophenolate Sodium (EC-MPS) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
C-reactive protein increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine (N=15) | Enteric-Coated Mycophenolate Sodium (EC-MPS) (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 4 | 4
Pyrexia (General disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Alveolar osteitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1
Ear infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Renal cyst infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure Restriction Description: The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.